CLINICAL TRIAL: NCT03879226
Title: Effects of Photobiomodulation Therapy in Aerobic Training and Detraining in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1781602-2
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Aerobic Endurance
Keywords: Photobiomodulation Therapy; Low-level Laser Therapy; Aerobic Endurance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher will program the device (placebo or PMBT) and will be instructed not to inform the volunteers or other researchers as to the type of treatment (PMBT or placebo). Therefore, the researcher responsible for the treatment will be blinded to the type of treatment being administered to the volunteers. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (placebo or PBMT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PBMT + training/ PBMT + detraining (Experimental): PBMT applied before and after the aerobic training sessions (12 weeks, 3 times a week) and PBMT applied during the detraining period (4 weeks, 3 times a week).
  Interventions: Device: PBMT
- PBMT + training/ placebo + detraining (Experimental): PBMT applied before and after the aerobic training sessions (12 weeks, 3 times a week) and placebo applied during the detraining period (4 weeks, 3 times a week).
  Interventions: Device: PBMT; Device: Placebo
- Placebo + training/ PBMT + detraining (Experimental): Placebo applied before and after the aerobic training sessions (12 weeks, 3 times a week) and PBMT applied during the detraining period (4 weeks, 3 times a week).
  Interventions: Device: PBMT; Device: Placebo
- Placebo + training/ placebo + detraining (Placebo Comparator): Placebo applied before and after the aerobic training sessions (12 weeks, 3 times a week) and placebo applied during the detraining period (4 weeks, 3 times a week).
  Interventions: Device: Placebo

INTERVENTIONS:
Device: PBMT — PBMT will be applied bilaterally using the direct contact method with light pressure on the skin at different sites, namely 9 sites on the knee extensor muscles, 6 sites on the knee flexor muscles, and 2 sites on the plantar flexor muscles. A 12-diode cluster, with 4 905-nm laser diodes (12.5W peak power for each diode), 4 875-nm LED diodes (17.5 mW mean power for each diode), and 4 640-nm LED diodes (15 mW mean power for each diode), manufactured by Multi Radiance Medical® (Solon, OH, USA), will be used to apply the PBMT. The dose used for the applications during the training and/or detraining periods will be 30 Joules (J) per site (510 J per lower limb). PBMT will be applied before and after each training session and during the detraining period, depending on the group to which the volunteers are allocated.
  Arms: PBMT + training/ PBMT + detraining; PBMT + training/ placebo + detraining; Placebo + training/ PBMT + detraining
Device: Placebo — Placebo will be applied bilaterally using the direct contact method with light pressure on the skin at different sites, namely 9 sites on the knee extensor muscles, 6 sites on the knee flexor muscles, and 2 sites on the plantar flexor muscles. The placebo PBMT will per performed using the dose of 0 J per diode. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (active or placebo). Placebo will be applied before and after each training session and during the detraining period, depending on the group to which the volunteers are allocated.
  Arms: PBMT + training/ placebo + detraining; Placebo + training/ PBMT + detraining; Placebo + training/ placebo + detraining

SUMMARY:
In last years it has been demonstrated that photobiomodulation therapy (PBMT) has ergogenic effects. However some key aspects, such as the potentially beneficial effects of PBMT during the detraining period still remain unknown.

Therefore, the aim of this project is to evaluate the effects of PBMT applied before and after aerobic training sessions and during the detraining period.

DETAILED DESCRIPTION:
It will be carried out a randomized, triple-blind, placebo-controlled trial.

Seventy-two volunteers will be randomly allocated to four experimental groups:

1. PBMT before and after the aerobic training sessions and PBMT during the detraining period;
2. PBMT before and after the aerobic training sessions and placebo during the detraining period;
3. Placebo before and after the aerobic training sessions and PBMT during the detraining period;
4. Placebo before and after the aerobic training sessions and placebo during the detraining period .

The individuals randomly allocated to the different groups will be subjected to 12 consecutive weeks of aerobic training performed on a treadmill 3 times a week on non-consecutive days. Each training session will last 30 minutes, with an intensity ranging from 85 to 90% maximum heart rate. PBMT or placebo will be applied before and after each training session. After the 12-week training period, the volunteers will receive the application of PBMT or placebo depending on the group to which they are allocated for 4 weeks (3 times a week) without training.

The data will be collected by a blind assessor. It will be analyzed time of the exercise (time until exhaustion), maximum oxygen consumption in absolute and relative values in relation to body mass (VO2max). Moreover, it will be evaluated the body composition. The evaluations will be performed before starting the protocol (baseline) and after 4, 8, and 12 weeks of training. They will also be performed after 4 weeks without training (detraining period).

The findings will be tested for their normality using the Shapiro-Wilk test. Parametric data will be expressed as mean and standard deviation and nonparametric data as median and respective upper and lower limits. Parametric data will be analyzed by two-way repeated measures analysis of variance (ANOVA; time versus experimental group) with post-hoc Bonferroni correction. Non-parametric data will be analyzed using the Friedman test and, secondarily, the Wilcoxon signed-rank test. Data will be analyzed in terms of both their absolute values and their relationship to the percentage change based on the values established in the baseline tests. The significance level will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men;
* Aged from 18 to 35 years;
* Complete at least 80% of the study procedures will be included in the study.

Exclusion Criteria:

* History of musculoskeletal injury in the hip and knee regions in the 2 months before the study;
* Become injured during the study;
* Regularly use pharmacological agents and/ or nutritional supplements;
* Signs and symptoms of any neurological, metabolic, inflammatory, pulmonary, oncological, or cardiovascular disease that may limit the execution of high-intensity exercises.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2019-08-25 (Actual)

PRIMARY OUTCOMES:
Time until exhaustion. | 16 weeks - 4 weeks after completing the training (detraining period).
  The time until exhaustion will be measured by the software of ergospirometry system.

SECONDARY OUTCOMES:
Time until exhaustion. | 4, 8, and 12 weeks after starting the training period.
  The time until exhaustion will be measured by the software of ergospirometry system.
Maximum oxygen consumption (VO2). | 4, 8, and 12 weeks after starting the training period, and at 4 weeks after completing the training (detraining period).
  The rates of maximum oxygen consumption will be measured by an ergospirometry test.
Fat percentage. | 4, 8, and 12 weeks after starting the training period, and at 4 weeks after completing the training (detraining period).
  Fat percentage will be measured by diameters, perimeters, and skinfolds.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar Pinto Leal Junior, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request addressed to the principal investigator.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] de Paiva PRV, Casalechi HL, Tomazoni SS, Machado CDSM, Ribeiro NF, Pereira AL, de Oliveira MFD, Alves MNDS, Dos Santos MC, Takara IET, Miranda EF, de Carvalho PTC, Leal-Junior ECP. Does the combination of photobiomodulation therapy (PBMT) and static magnetic fields (sMF) potentiate the effects of aerobic endurance training and decrease the loss of performance during detraining? A randomised, triple-blinded, placebo-controlled trial. BMC Sports Sci Med Rehabil. 2020 Apr 10;12:23. doi: 10.1186/s13102-020-00171-2. eCollection 2020. PMID 32308987
- [Derived] de Paiva PRV, Casalechi HL, Tomazoni SS, Machado CDSM, Miranda EF, Ribeiro NF, Pereira AL, da Costa AS, Dias LB, Souza BCG, Aguiar Lino MM, de Carvalho PTC, Leal-Junior ECP. Effects of photobiomodulation therapy in aerobic endurance training and detraining in humans: Protocol for a randomized placebo-controlled trial. Medicine (Baltimore). 2019 May;98(18):e15317. doi: 10.1097/MD.0000000000015317. PMID 31045769